CLINICAL TRIAL: NCT04714840
Title: Telehealth Based Intervention to Improve Functional Capacity in Survivors of Childhood Cancer With Significantly Limited Exercise Tolerance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CARTOXIII; U01CA246570-01 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2021-01-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer; Mobility Limitation
MeSH Terms: conditions — Neoplasms; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized exercise group (INTGroup) (Other): Participants in this group have individually tailored exercise program with supervision, 20 weeks,clinic 3 times during the course of this study: at baseline (this appointment), at 4 months and 10 months from now for follow-up.
  Interventions: Other: Exercise testing results; Other: Individually tailored exercise program (INT)
- Generalized exercise group, Attention Control (AC Group) (Other): Study participants in this group receive generalized exercise recommendations, 20 weeks,clinic 3 times during the course of this study: at baseline (this appointment), at 4 months and 10 months from now for follow-up.
  Interventions: Other: Exercise testing results; Other: Generalized exercise recommendations (AC)

INTERVENTIONS:
Other: Exercise testing results — Tailored, home-delivered aerobic and strengthening intervention,exercise intolerance,Both groups of participants will be provided with the results of their exercise testing.
Other: Individually tailored exercise program (INT) — Individuals randomized to receive an individually tailored exercise program will meet with an exercise specialist. Written instructions, videos of each strengthening exercise, a blue tooth enable heart rate monitor, all necessary exercise equipment, and an iPad pre-loaded with heart rate monitor software, exercise videos and ZOOM app (for video conferencing) will be provided. After returning home, the exercise specialist will supervise and provide guidance to the individual via the ZOOM app during the first 2 weeks (3 sessions per week). Supervision will slowly decrease to twice a week in weeks 3-4, once a week in weeks 5-8, every other week in weeks 9-16, and to one time midway between weeks 17-20. The exercise program will be adjusted depending on the individuals progress.
  Arms: Personalized exercise group (INTGroup)
Other: Generalized exercise recommendations (AC) — Individuals randomized to receive the generalized exercise recommendations will receive a copy of the Physical Activity Guidelines for Americans. At the baseline visit, a study staff will review these guidelines and answer questions about their exercise testing and encourage them to be physically active. The staff will contact them via telephone to complete a short questionnaire weekly during weeks 1-8 and monthly for weeks 9-20.
  Arms: Generalized exercise group, Attention Control (AC Group)

SUMMARY:
The participants are asked to take part in this clinical trial, a type of research study. The participants are SJLIFE study participants and may have a hard time exercising (exercise intolerance) due to side effects of cancer treatment received as a child.This study is being done to determine if a personalized exercise plan will help childhood cancer survivors who have exercise intolerance become more active.

Primary Objectives:

To achieve the goal of this study, we propose the following three Objectives:

Primary Objective 1:

To determine the efficacy of an individually tailored, home-delivered aerobic and strengthening intervention to improve exercise capacity in survivors of childhood cancer with exercise intolerance (peak oxygen uptake (peak VO2) <85% of age and sex predicted).

Primary Objective 2:

To determine the effects of an individually tailored, home-delivered aerobic and strengthening intervention on measures of cardiac, pulmonary, musculoskeletal, and neurosensory function in survivors of childhood cancer with exercise intolerance.

Primary Objective 3:

To determine the effects of an individually tailored, home-delivered aerobic and strengthening intervention on emotional health, participation in family and community activities, quality of life, and cognitive function in survivors of childhood cancer with exercise intolerance.

DETAILED DESCRIPTION:
The design for this study will be a single-blind two-arm, prospective, randomized clinical trial. Performance testing results: Both groups of participants will be provided with the results of their performance testing. Individually tailored exercise program: Individuals randomized to receive an individually tailored exercise program will meet with an exercise specialist.Generalized exercise recommendations: Individuals randomized to receive the generalized exercise recommendations will receive a copy of the Physical Activity Guidelines for Americans.

ELIGIBILITY:
Inclusion Criteria:

* Between 18.00 and 39.99 years of age at the time of enrollment
* SJLIFE participant
* Peak VO2 <85% predicted
* Verbalizes understanding of directions for use of ZOOM on the study provided iPad and heart rate monitor
* Clearance for participation in exercise by a study physician
* Internet access

Exclusion Criteria:

* Enrolled in a formal exercise intervention
* Self-report of engaging in > 150 minutes/week of moderate physical activity
* Currently pregnant (assess by urine pregnancy test)
* Significant psychological distress (e.g. suicidal ideation)
* Requires immediate medical intervention (e.g. angina, decompensated heart failure)
* Research Participant Recruitment and Screening

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | Baseline to Week 20
  Changes in Peak VO2/2-minute step in place test in both INT and AC groups
Exercise capacity | Week 20 to 6 months after week 20
  Sustainability of changes in Peak VO2/2-minute step in place test in both INT and AC groups

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | baseline, week 20, 6 months after week 20
  Scale: 4 Options - Not at all (minimum value = 0), Several days (1), More than half the days (2), Nearly every day (maximum value = 3). Higher score = worse outcome. Possible score range is 0-27.
Generalized Anxiety Disorder (GAD-7) | baseline, week 20, 6 months after week 20
  Scale: 5 Options - Not at all sure (minimum value = 0), Several days (1), Over half the days (2), Nearly every day (maximum value = 3). Higher score = worse outcome. Possible score range is 0-21.
PROMIS Ability to Participate 8a (SF v2.0) | baseline, week 20, 6 months after week 20
  Scale: 5 Options - Never (maximum value = 5), Rarely (4), Sometimes (3), Usually (2), Always (minimum value = 1). Higher score = better outcome. Possible score range 8-40.
Work Productivity and Activity Impairment Questionnaire (WPAI) | baseline, week 20, 6 months after week 20
  Scale doesn't apply to overall questionnaire. Outcomes are expressed as impairment percentages. Higher numbers = worse outcome.
Work and Social Adjustment Scale (WSAS) | baseline, week 20, 6 months after week 20
  Scale: 0-8; Not at all (minimum value = 0) to Very Severely (maximum value = 8). Higher score = worse outcome. Possible score range 0-40.
Medical Outcomes Survey Short Form (SF-36) | baseline, week 20, 6 months after week 20
  Consists of 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Higher score = better outcome.
Childhood Cancer Survivor Study Neurocognitive Questionnaire - Revised (CCSS-NCQ) | baseline, week 20, 6 months after week 20
  Scale: 3 Options - Never a Problem (maximum value = 2), Sometimes a Problem (1) , Often a Problem (minimum value = 0). Higher score = better outcome. Possible score range 0-64.
PROMIS Global Health Short Forms | weekly during the first eight weeks and every four weeks during weeks 9-20
  brief global physical and mental health questionnaires; Scale: 5-point Likert scale, Excellent=5, Poor=1

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Ness, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- [Derived] Maharaj A, Jefferies JL, Mulrooney DA, Armstrong GT, Brinkman TM, O'Neil ST, Terrell S, Partin RE, Srivastava DK, Hudson MM, Wang Z, Ness KK. Design and methods of a randomized telehealth-based intervention to improve fitness in survivors of childhood cancer with exercise intolerance. Contemp Clin Trials. 2023 Oct;133:107339. doi: 10.1016/j.cct.2023.107339. Epub 2023 Sep 18. PMID 37730199
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04714840/ICF_000.pdf